CLINICAL TRIAL: NCT04849260
Title: Phase Ib/II, Open Label, Controlled Clinical Study of Pexa-Vec (Vaccinia GM CSF / Thymidine Kinase-Deactivated Virus) Combined With Recombinant Whole Human Anti-PD-L1 Monoclonal Antibody (ZKAB001) in Metastatic Melanoma After First-line Treatment Failure
Brief Title: Phase Ib/II Clinical Study of Pexa-Vec (Vaccinia GM CSF / Thymidine Kinase-Deactivated Virus) Combined With Recombinant Whole Human Anti-PD-L1 Monoclonal Antibody (ZKAB001) in Metastatic Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKAB001-LEES-2019-02
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Local Progression or Metastatic Melanoma With Failed First-line Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pexa-Vec combined with ZKAB001 (Experimental): The combined treatment group is divided into two dose groups. The principle of "3+3" is adopted to determine RP2D, and RP2D will be used in subsequent patients in this cohort.
  Interventions: Biological: Pexa-Vec combined with ZKAB001
- ZKAB001 monotherapy (Active Comparator): ZKAB001 monotherapy.
  Interventions: Biological: ZKAB001 monotherapy

INTERVENTIONS:
Biological: Pexa-Vec combined with ZKAB001 — 1. Intratumoral injection of low dose Pexa-Vec (3×10^8pfu) combined with intravenous of ZKAB001 (5mg/kg), every 2 weeks as one cycle.
  2. Intratumoral injection of high dose Pexa-Vec (1×10^9pfu) combined with intravenous of ZKAB001 (5mg/kg), every 2 weeks as one cycle.
  Arms: Pexa-Vec combined with ZKAB001
Biological: ZKAB001 monotherapy — ZKAB001 monotherapy
  Arms: ZKAB001 monotherapy

SUMMARY:
The study will be divided into two stages: phase Ib and phase II. The safety and phase II recommended dose (RP2D) of Pexa-Vec combined with ZKAB001 in patients with local progression of failed first-line treatment or metastatic melanoma will be evaluated in phase Ib.

Objective response rate (ORR) and progression-free survival (PFS) of ZKAB001 combined with RP2D's Pexa-Vec or ZKAB001 monotherapy in patients with local progression or metastatic melanoma will be evaluated in phase II.

DETAILED DESCRIPTION:
The study will be divided into two stages: phase Ib and phase II. The safety and phase II recommended dose (RP2D) of Pexa-Vec combined with ZKAB001 in patients with local progression of failed first-line treatment or metastatic melanoma will be evaluated in phase Ib.

Objective response rate (ORR) and progression-free survival (PFS) of ZKAB001 combined with RP2D's Pexa-Vec or ZKAB001 monotherapy in patients with local progression or metastatic melanoma will be evaluated in phase II.

The study is also going to evaluate the combination therapy or monotherapy:

1. overall survival time ((OS)), disease control rate (DCR) and duration of remission (DOR) in patients with metastatic melanoma.
2. safety
3. the relationship between the expression of PD-L1 in tumor tissue and clinical effect；
4. the changes of immune microenvironment (CD8+ expression) in tumor tissue before and after Pexa-vec treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent.
2. Age 18-75 years old (inclusive), regardless of gender.
3. Pathologically proved to be malignant melanoma, including skin, mucous membrane, and limb origin, and locally progressive or metastatic melanoma that cannot be completely resected.
4. The patient has more than 1 superficial focus for intratumoral injection (suitable for direct or ultrasound-guided injection), which can be skin, subcutaneous or lymph node focus, the longest diameter is (LD) ≥ 1cm and ≤ 10cm, and there is no ulcer in the injected focus.
5. Patients who have failed to receive first-line treatment of melanoma in the past, including chemotherapy and targeted therapy.

   Systemic anticancer therapy or adjuvant therapy must be completed at least 4 weeks before enrollment (if previously received nitrosourea or mitomycin C chemotherapy, the interval between the end of chemotherapy and the study group is more than 6 weeks).

   Patients with adverse events caused by previous treatment recovered to ≤ CTCAE level 1, except for hair loss.
6. Measurable lesions based on RECISTv 1.1.
7. The ECOG physical condition score is 0 or 1, and the expected survival time is more than 3 months.
8. The functions of blood, liver and kidney are good and meet the results of laboratory tests:

1) Absolute neutrophil count (ANC) ≥ 1.5x10^9 / L. 2) Platelet ≥ 80 × 10^9 shock L. 3) Hemoglobin ≥ 90g/L. 4) Serum albumin ≥ 28g/L. 5) Bilirubin ≤ 1.5x ULN. 6) ALT and AST ≤ 2.5x ULN, if there is liver metastasis, ALT and AST ≤ 5x ULN. 7) Serum Cr ≤ 1.25 × ULN or endogenous creatinine clearance ≥ 50mL/min (using standard Cockcroft-Gault formula).

8) Coagulation function, in which INR ≤1.5 ULN. 9. Female or male patients of childbearing age should take effective contraceptive methods during the study period and within 3 months after the end of the study treatment period. Non-operative sterilization female patients of childbearing age must be negative for serum HCG test during the screening period.

Exclusion Criteria:

1. Active, known or suspected autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granuloma, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis.

   Residual hypothyroidism caused by autoimmune thyroiditis that only requires hormone replacement therapy, controlled type I diabetes, or the absence of external stimulation that is not expected to recur can be included. Patients with eczema, psoriasis, neurodermatitis or vitiligo (patients with psoriatic arthritis will need to be excluded) who only have skin symptoms can be enrolled in the group if they meet the following conditions: the area covered by the rash must be less than 10% of the body surface area; the disease is well controlled at the baseline level, requiring only local steroids, and those with no acute exacerbation in the past 12 months can be included.
2. Subjects were treated with immunosuppressants or systemic or absorbable local corticosteroids within 2 weeks before enrollment to achieve immunosuppression (dose > 10mg/ prednisone or equivalent).
3. Has received or plans to receive any form of organ transplant, including allogeneic stem cell transplantation.
4. Known to be allergic to macromolecular protein preparations, or to any composition of ZKAB001 and Pexa-Vec.
5. Severe allergic reactions or side effects occurred in the past vaccination process.
6. Complications of other malignant tumors less than 5 years before the first dose, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, ductal carcinoma in situ after radical resection (hormone therapy for non-metastatic prostate cancer or breast cancer is acceptable)
7. Subjects with known active central nervous system (CNS) metastasis and / or carcinomatous meningitis.

   Note: subjects who have previously received brain metastasis treatment and subjects with clinically stable CNS metastasis may be allowed to participate in the study (defined as at least 4 weeks before the first dose of the trial treatment: (1) No new or expanded evidence of CNS metastasis (through MRI); (2) subjects have been treated without hormones for at least 2 weeks; (3) any neurological symptoms have returned to baseline levels.
8. Patients with uncontrolled cardiac clinical symptoms or diseases, such as heart failure above NYHA2, unstable angina pectoris, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, left ventricular ejection fraction at rest was less than 50%.
9. After injection treatment, tumor swelling and / or necrosis may invade important vascular structures (such as carotid artery) or other important anatomical sites (such as spinal cord).
10. A history of severe inflammatory skin diseases requiring drug treatment and a history of severe eczema requiring drug treatment (confirmed by researchers).
11. The subjects had active infection, or had a fever of unknown origin during the screening period or within a week before the first administration of the drug > 38.5 ℃. (according to the judgment of the researchers, the fever caused by the tumor can be included in the group.).
12. Active hepatitis B or C (unless HBV-DNA titer < 500IU/mL or copy number < 1000copies/ml, HCV-RNA negative can be included in), HIV positive or known history of acquired immunodeficiency syndrome after antiviral treatment.
13. Subjects are participating in other clinical studies, or less than one month from the end of the previous clinical study, except for non-interventional clinical studies (such as epidemiological studies).
14. HCV therapy could not be stopped within 14 days before Pexa-Vec injection. If a patient is using any antiviral drugs, he or she should consult the researcher to determine whether the patient is suitable to participate in the study.
15. Less than 4 weeks from the previous use of immune checkpoint inhibitors, such as PD-1/CTLA-4 inhibitors (that is, more than 4 weeks from the previous receipt of PD-1/CTLA-4 inhibitors); or have been treated with other oncolytic viruses (such as T-Vec, recombinant human GM-CSF herpes simplex virus injection (OrienX010), etc.) or PD-L1 inhibitors.
16. The patients were vaccinated with live vaccine within 4 weeks before screening. Inactivated vaccines to prevent influenza and inactivated vaccines to prevent other infectious diseases can be used on a case-by-case basis, but it is necessary to consider increasing the elution period before and after medication.
17. Subjects are known to have a history of psychotropic substance abuse, alcohol abuse or drug use.
18. Subjects with active pulmonary tuberculosis or with a history of active pulmonary tuberculosis infection within 1 year before medication, with or without treatment.
19. The researchers evaluated that there was a significant bleeding event in the previous 12 months and the risk of intratumoral injection procedure increased.
20. Pregnant or lactating women.
21. The researchers determined that the patient had other factors that might lead to the termination of the study, such as other serious diseases or serious laboratory abnormalities or accompanied by other factors that would affect the safety of the subjects, or family or social factors such as the collection of trial data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
dose-limited toxicity (DLT) | 28 days after first dose
  dose-limited toxicity (DLT)
maximum tolerated dose (MTD) | 28 days after first dose
  recommended phase 2 dose RP2D.
progression free survival (PFS) | 2 years
  progression free survival
objective response rate | 2 years
  objective response rate

SECONDARY OUTCOMES:
disease control rate (DCR) | 2 years
  disease control rate
duration of response (DOR) | 2 years
  duration of response
6-month and 1-year PFS rate | 12 months
  6-month and 1-year PFS rate
1-year and 2-year OS rates | 2 years
  1-year and 2-year OS rates
AE/SAEs | 2 years
  The incidence and severity of adverse events (AE) and severe adverse events (SAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No